CLINICAL TRIAL: NCT00240708
Title: A Parallel-Group Comparative Open-Label Study of Long-Acting Injectible Risperidone Versus Risperidone Tablets in Patients With Schizophrenia.
Brief Title: A Study of the Efficacy and Safety of Long-acting Injectable Risperidone and Risperidone Tablets in Patients With Schizophrenia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Janssen Pharmaceutical K.K. (Industry)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CR004945
Record Dates: First submitted 2005-10-14; First posted 2005-10-18 (Estimated); Last update posted 2011-05-17 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; intramuscular injection; antipsychotic agents; risperidone; long-acting injectable
MeSH Terms: conditions — Schizophrenia | interventions — Risperidone

INTERVENTIONS:
Drug: risperidone

SUMMARY:
The purpose of this study is to evaluate the effectiveness and safety of risperidone, formulated as a long-acting injectable drug, compared with risperidone tablets in the treatment of patients with schizophrenia.

DETAILED DESCRIPTION:
Although many schizophrenia patients currently take oral antipsychotic medications, it is estimated that up to 75% of them have difficulty adhering to the daily oral regimen. Long-acting injectable formulations may eliminate the need for daily medication and enhance patient compliance with the treatment regimen. This is an open-label, randomized, Phase III trial in patients with schizophrenia. One treatment group receives 25 to 50 mgs of long-acting risperidone, formulated for intramuscular injections, at study initiation and again after 2 weeks, while phasing out any previous antipsychotic medication during the initial 3 weeks of the study. Continuing in the treatment phase, long-acting injections are administered once every 2 weeks through Week 24, and post-treatment observation is performed for 6 weeks (total study duration of 30 weeks). Patients in the other treatment group take oral risperidone tablets, 2 to 6 mgs daily, from study initiation for 24 weeks. Post-treatment observation continues for 1 week for this group (total study duration of 25 weeks). Assessments of effectiveness made at specified intervals during treatment include Positive And Negative Syndrome Scale (PANSS), a scale for the measurement of symptoms of schizophrenia; Clinical Global Impression - Severity (CGI-S), a measure of overall severity of illness, and Clinical Global Impression - Changes (CGI-C); as well as, Brief Psychiatric Rating Scale (BPRS). Safety evaluations include the incidence of adverse events throughout the study; inspection of the injection site at times of treatment; Drug-Induced Extrapyramidal Symptoms Scale (DIEPSS), vital signs (pulse, blood pressure, temperature), and laboratory tests (hematology, biochemistry, urinalysis) at monthly intervals. The study hypothesis is that treatment with long-acting risperidone injections is not inferior to oral risperidone, as measured by changes in PANSS total score from baseline through endpoint (24 weeks), in patients with schizophrenia and is generally well-tolerated. Risperidone, long-acting formulation for intramuscular injections (25 milligrams[mg] to 50mg, maximum), given biweekly through 24 weeks. Oral risperidone (2mg/day to 6mg/day [maximum]) administered daily for 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of schizophrenia by the criteria of Diagnostic and Statistical Manual of Mental Diseases, 4th Edition (DSM-IV )
* treatment with an antipsychotic drug (up to 6 milligrams/day of risperidone or equivalent dose) for 28 days before study initiation with no change in the dosage
* Total Positive and Negative Syndrome Scale (PANSS) score >=60 and <120 at start of study.

Exclusion Criteria:

* Diagnosis of mental disease other than schizophrenia
* treated with a sustained-release injection of other antipsychotic medications within 60 days before the initiation of the study
* history of cerebrovascular accident, convulsive disorder such as epilepsy, diabetes mellitus, liver disease, kidney disease, cardiovascular disorder, malignancy or physical exhaustion due to dehydration or malnutrition
* have risk factors of diabetes mellitus, such as hyperglycemia.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2004-06; Study Completion 2006-04 (Actual)

PRIMARY OUTCOMES:
Positive and Negative Syndrome Scale (PANSS) at screening, Weeks 8, 16, and 24.

SECONDARY OUTCOMES:
Clinical Global Impression-Changes (CGI-C), from baseline at Weeks 8, 16 and 24; Brief Psychiatric Rating Scale (BPRS) at baseline and biweekly from Weeks 4 through 18; Clinical Global Impressions-severity (CGI-S)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Pharmaceutical K.K. Clinical Trial, Study Director — Janssen Pharmaceutical K.K.

REFERENCES:
- [Derived] Ostuzzi G, Bighelli I, So R, Furukawa TA, Barbui C. Does formulation matter? A systematic review and meta-analysis of oral versus long-acting antipsychotic studies. Schizophr Res. 2017 May;183:10-21. doi: 10.1016/j.schres.2016.11.010. Epub 2016 Nov 17. PMID 27866695
- See also: A study of the Efficacy and Safety of Long-Acting injectible Risperidone and Risperidone tablets in patients with Schizophrenia. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=409&filename=CR004945_CSR.pdf